CLINICAL TRIAL: NCT02722928
Title: Impact of Intraoperative Ventilation With High Oxygen Content to Reduce the Incidence and Extent of Postoperative Pneumocephalus in Patients Undergoing Craniotomies
Brief Title: Ventilation With High Oxygen Content and Postoperative Pneumocephalus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Variability of the pneumocephalus volume mean was higher than initially assumed
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Gurneet Sandhu, M.D., Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2015H0032
Record Dates: First submitted 2016-03-21; First posted 2016-03-30 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Pneumocephalus
Keywords: Postoperative pneumocephalus; Fraction of inspired oxygen; Intracranial surgery
MeSH Terms: conditions — Pneumocephalus | interventions — Oxygen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional 1:1 oxygen/air gas mixture (No Intervention): 80 patients will receive ventilation during the surgery with a 1:1 oxygen / air gas mixture
- Pure oxygen ventilation (Experimental): Patients will receive controlled ventilation with a conventional 1:1 oxygen / air gas mixture (60% oxygen concentration) during the approach and tumor removal phases. Once tumor resection is completed and hemostasis started, this group of patients will be switched to ventilation with 100% (pure) oxygen concentration
  Interventions: Other: Controlled Ventilation with 100% oxygen

INTERVENTIONS:
Other: Controlled Ventilation with 100% oxygen — Patients in group B will be switched from conventional 1:1 oxygen / air ventilation to 100% oxygen controlled ventilation once tumor resection is completed and hemostasis started. They will inhale 100% oxygen until extubation
  Other Names: FiO2 100% after tumor resection
  Arms: Pure oxygen ventilation

SUMMARY:
The aim of this study is to compare the incidence and volume of postoperative pneumocephalus in patients receiving ventilation with 100% oxygen during the last stage of surgery versus a conventional 1:1 oxygen/air gas mixture.

DETAILED DESCRIPTION:
Background: Postoperative pneumocephalus is a common complication in patients undergoing craniotomies. Even though the treatment of postoperative pneumocephalus with the use of supplemental oxygen is well documented, yet not reports have shown its role for the prevention of this condition. We suggest the use of intraoperative ventilation with 100% oxygen as prophylaxis for the incidence and severity of postoperative pneumocephalus in patients undergoing intracranial surgery.

Objectives: The aim of this study is to compare the incidence and volume of postoperative pneumocephalus in patients receiving ventilation with 100% oxygen during the last stage of surgery versus a conventional 1:1 oxygen/air gas mixture.

Study Methods: A single-blinded, prospective study, randomizing 80 patients per group, expecting 80% power to detect a 20% decrease in pneumocephalus volume for the interventional group. Inclusion criteria: Patients >18 years, scheduled to undergo elective craniotomy, and be willing to give written informed consent.

Study Procedures: Once the tumor resection is completed and hemostasis started (beginning of stage 2), patients will be assigned to receive either 1:1 oxygen/air gas mixture (control group) or 100% oxygen (intervention group) until the end of the surgery. All patients will receive postoperative supplemental oxygen via nasal cannula. CT scan will be performed within 1 to 6 postoperative hours as standard of care. A blinded radiologist will review all CT scans and assess the extent and frequency of postoperative pneumocephalus.

Clinical Outcomes: Patients' demographic data, length of stage 2, period of time between the end of surgery and CT scan, and pneumocephalus volumetric measurements will be compared between groups. Baseline neurological status will be compared with clinical and imaging postoperative findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of both sexes undergoing surgical procedures to treat hemispheric or posterior cranial fossa tumors and consenting to the study

Exclusion Criteria:

* History of severe cardio-pulmonary disease.
* Bleeding disorders
* Previous neurosurgeries requiring cranial reconstruction
* Head trauma
* Decreased consciousness related to cerebral edema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08; Primary Completion 2018-01 (Actual); Study Completion 2018-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gurneet Sandhu, M.D., Principal Investigator — Ohio State University
Locations (1):
- Department of Anesthesiology - Clinical Research, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beppu T, Ogasawara K, Ogawa A. Alleviation of intracranial air using carbon dioxide gas during intraventricular tumor resection. Clin Neurol Neurosurg. 2006 Oct;108(7):655-60. doi: 10.1016/j.clineuro.2006.01.002. Epub 2006 Feb 14. PMID 16483713
- [Background] Schirmer CM, Heilman CB, Bhardwaj A. Pneumocephalus: case illustrations and review. Neurocrit Care. 2010 Aug;13(1):152-8. doi: 10.1007/s12028-010-9363-0. PMID 20405340
- [Background] Gore PA, Maan H, Chang S, Pitt AM, Spetzler RF, Nakaji P. Normobaric oxygen therapy strategies in the treatment of postcraniotomy pneumocephalus. J Neurosurg. 2008 May;108(5):926-9. doi: 10.3171/JNS/2008/108/5/0926. PMID 18447708
- [Background] Aoki N, Sakai T. Computed tomography features immediately after replacement of haematoma with oxygen through percutaneous subdural tapping for the treatment of chronic subdural haematoma in adults. Acta Neurochir (Wien). 1993;120(1-2):44-6. doi: 10.1007/BF02001468. PMID 8434516
- [Background] Branger AB, Lambertsen CJ, Eckmann DM. Cerebral gas embolism absorption during hyperbaric therapy: theory. J Appl Physiol (1985). 2001 Feb;90(2):593-600. doi: 10.1152/jappl.2001.90.2.593. PMID 11160058
- [Derived] Sandhu G, Gonzalez-Zacarias A, Fiorda-Diaz J, Soghomonyan S, Abdel-Rasoul M, Prevedello LM, Uribe AA, Stoicea N, Targonski D, Prevedello DM, Bergese SD. A prospective randomized clinical trial to evaluate the impact of intraoperative ventilation with high oxygen content on the extent of postoperative pneumocephalus in patients undergoing craniotomies. Br J Neurosurg. 2019 Apr;33(2):119-124. doi: 10.1080/02688697.2018.1562031. Epub 2019 Feb 20. PMID 30784332

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional 1:1 Oxygen/Air Gas Mixture: 39 patients received ventilation during the surgery with a 1:1 oxygen / air gas mixture
- Pure Oxygen Ventilation: 31 patients received controlled ventilation with a conventional 1:1 oxygen / air gas mixture during the approach and tumor removal phases. Once tumor resection was completed and hemostasis started, this group of patients was switched to ventilation with pure oxygen (FiO2 = 100%) until extubation
Period: Overall Study
Arm/Group | Conventional 1:1 Oxygen/Air Gas Mixture | Pure Oxygen Ventilation
Started | 49 | 51
Completed | 39 | 31
Not Completed | 10 | 20
Not completed — Standard CT was not as required per prot | 5 | 13
Not completed — Required Intraoperative MRI | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional 1:1 Oxygen/Air Gas Mixture | Pure Oxygen Ventilation | Total
Number analyzed (Participants) | 39 | 31 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.69 (14.21) | 50.81 (13.28) | 48.51 (13.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 14 | 37
  Male | 16 | 17 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 36 | 27 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 31 | 70
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 31.35 (7.42) | 31.94 (6.64) | 31.61 (7.04)
American Society of Anesthesiologists Physical Status (ASA PS) [Count of Participants; unit: Participants] — ASA PS classification describes the preoperative clinical status of the patient. ASA PS comprise 6 levels. The last 2 (ASA PS V and VI) are for moribund and brain death patients respectively and therefore, were not included in our patient setting. The following categories were included in our trial: ASA PS I: A normal healthy patient; ASA PS II: A patient with mild systemic disease; ASA PS III: A patient with severe systemic disease; ASA PS IV: A patient with severe systemic disease that is a constant threat to life
  Participants
    ASA PS I | 0 | 1 | 1
    ASA PS II | 12 | 9 | 21
    ASA PS III | 26 | 20 | 46
    ASA PS IV | 1 | 1 | 2
Preoperative Diagnosis [Count of Participants; unit: Participants] — Supratentorial lesions are the ones located above the tentorium cerebelli (e.g. cerebral lesions) Infratentorial lesions are the ones located below the tentorium cerebelli (e.g. cerebellar lesions)
  Participants
    Supratentorial Lesion (above tentorium cerebelli) | 25 | 21 | 46
    Infratentorial Lesion (below tentorium cerebelli) | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Volume of Postoperative Pneumocephalus
Description: Compare the extent (cm3) of postoperative pneumocephalus in patients ventilated intraoperatively with 100% oxygen during hemostasis and wound closure versus 1:1 oxygen / air mixture
Time Frame: One to six hours after surgery
Measure: Median (Inter-Quartile Range); unit: cm^3
Arm/Group | Conventional 1:1 Oxygen/Air Gas Mixture | Pure Oxygen Ventilation
Number analyzed (Participants) | 39 | 31
cm^3 | 9.65 [3.61 to 23.20] | 7.06 [2.70 to 20.1]

2. Primary Outcome: Occurrence of Postoperative Pneumocephalus
Description: Compare the occurrence rate of postoperative pneumocephalus (present or not present) in patients receiving intraoperative ventilation with 100% oxygen during hemostasis and wound closure versus 1:1 oxygen / air mixture
Time Frame: One to six hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional 1:1 Oxygen/Air Gas Mixture | Pure Oxygen Ventilation
Number analyzed (Participants) | 39 | 31
Participants | 39 | 31

3. Secondary Outcome: Pneumocephalus Volume and Anterior Fossa Surgery
Description: To compare the presence of postoperative pneumocephalus in patients who underwent anterior fossa surgery.
Time Frame: One to six hours after surgery
Measure: Median (Inter-Quartile Range); unit: cm^3
Groups:
- Conventional 1:1 Oxygen/Air Gas Mixture: Out of the 39 patients included in the Conventional 1:1 oxygen / air gas mixture ventilation group, 23 patients underwent conventional anterior fossa surgery. Pneumocephalus volume was compared between groups for this patient sub-setting
- Pure Oxygen Ventilation: Out of the 31 patients in the pure oxygen ventilation after hemostasis group, 16 patients underwent conventional anterior fossa surgery. Pneumocephalus volume was compared between groups for this patient setting
Arm/Group | Conventional 1:1 Oxygen/Air Gas Mixture | Pure Oxygen Ventilation
Number analyzed (Participants) | 23 | 16
cm^3 | 17.4 [6.89 to 24.4] | 13.95 [4.82 to 22.15]

4. Secondary Outcome: Pneumocephalus Volume and Posterior Fossa Surgery
Description: Pneumocephalus volume in patients who underwent posterior fossa surgery
Time Frame: one to six hours after surgery
Measure: Median (Inter-Quartile Range); unit: cm^3
Groups:
- Conventional 1:1 Oxygen / Air Gas Mixture Ventilation: Out of the 39 patients in the Conventional 1:1 oxygen / air gas mixture ventilation group, 15 patients underwent conventional posterior fossa surgery. Pneumocephalus volume was compared between groups for this patient sub-setting
- Pure Oxygen Ventilation After Hemostasis: Out of the 31 patients in the pure oxygen ventilation after hemostasis group,11 patients underwent conventional posterior fossa surgery. Pneumocephalus volume was compared between groups for this patient sub-setting
Arm/Group | Conventional 1:1 Oxygen / Air Gas Mixture Ventilation | Pure Oxygen Ventilation After Hemostasis
Number analyzed (Participants) | 15 | 11
cm^3 | 4.38 [0.81 to 10.50] | 4.00 [0.60 to 13.00]

5. Secondary Outcome: Changes in Neurological Outcomes at POD 3 Compared to Preoperative Evaluation
Description: Changes in Neurological Outcomes from baseline (preoperative evaluation) were documented based on differences (if any) found between both physical examinations: baseline (before surgery) and postoperative day (POD) 3 neurological exam. Results were reported as "improvement" (partial or total recovery of baseline neurological signs/symptoms), "no changes", and "deterioration" (focal or global neurological deterioration) in comparison with baseline neurological examination
Time Frame: preoperative to postoperative day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional 1:1 Oxygen/Air Gas Mixture | Pure Oxygen Ventilation
Number analyzed (Participants) | 39 | 31
Participants
  Improvement from baseline | 8 | 6
  No changes from baseline | 25 | 15
  Deterioration from baseline | 6 | 10

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the surgery start date / time to postoperative day 3
Groups:
- Pure Oxygen Ventilation: 31 patients received controlled ventilation with a conventional 1:1 oxygen / air gas mixture (60% oxygen concentration) during the approach and tumor removal phases. Once tumor resection was completed and hemostasis started, this group of patients was switched to ventilation with pure oxygen (100% oxygen concentration) until extubation
Arm/Group | Conventional 1:1 Oxygen/Air Gas Mixture | Pure Oxygen Ventilation
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/31
Other Adverse Events (participants affected / at risk) | 0/39 | 0/31

LIMITATIONS AND CAVEATS:
Sample size calculations were based on published data and resulted in the trial being under-powered. We did not incorporate a second postoperative CT scan to evaluate the changes in pneumocephalus volume during the immediate postoperative period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT02722928/Prot_SAP_000.pdf